CLINICAL TRIAL: NCT03519373
Title: Impact of HIV Infection and Pregnancy on Humoral Responses to Pertussis Immunization
Brief Title: Pertussis Immunization During Pregnancy & HIV Infection
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Principal Investigator, Nicolas Dauby, M.D. Ph.D., Centre Hospitalier Universitaire Saint Pierre
Other Study IDs: Pertussis
Record Dates: First submitted 2018-04-26; First posted 2018-05-09 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Immunization; Infection; Pertussis; HIV-1-infection; Pregnancy
MeSH Terms: conditions — Infections; Whooping Cough

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * PBMCs
  * Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- PER001: HIV 1-infected pregnant women
  Interventions: Biological: TDaP
- PER002: HIV 1-uninfected pregnant women
  Interventions: Biological: TDaP
- PER003: HIV 1-uninfected non-pregnant women
  Interventions: Biological: TDaP

INTERVENTIONS:
Biological: TDaP — Tetanus, Diphteria and Acellular Pertussis vaccine (Boostrix)

SUMMARY:
The impact of chronic HIV infection and pregnancy on different aspects of the humoral response to pertussis immunization with the TDaP vaccine will be studied. The parameters will be measured in 3 groups (HIV-infected pregnant, HIV-uninfected pregnant and HIV-uninfected non pregnant) at different time points before and after immunization (7-10 days, 30 days and at delivery). The transfer ratio and the quality of maternal antibodies will be studied in cord blood.

DETAILED DESCRIPTION:
Despite the growing importance of maternal immunization in the control of infectious pathogens in early life, the impact of pregnancy on vaccine immunogenicity remains poorly understood. Evidence suggests that pregnancy may influence the quality of the antibody response to vaccines. Pregnancy is associated with modifications in the glycosylation profile of immunoglobulins G (IgG). Different patterns of glycosylation are associated with differential regulation of the effector functions of IgG such as antibody-dependent cell cytotoxicity, complement activation or antibody dependent phagocytosis. Whether similar modifications affect vaccine-induced IgG in pregnant women is unknown.

HIV infection is associated with important alterations in B cells and antibodies. Although antiretroviral therapy partly corrects the proportions of memory B cells (MBC) subsets, it does not restore B cell responses to vaccines, measured as seroconversion rates and antibody persistence. Reduced IgG responses to vaccines have been observed in HIV-infected pregnant women but the impact of HIV on the quality of vaccine-induced IgG has not been reported. On the other hand, HIV infection in pregnancy has a strong impact on the transfer of maternal IgG to the newborn, possibly as a consequence of hypergammaglobulinemia and immune activation.

The investigators will:

1. Assess the respective impact of pregnancy and HIV infection on the magnitude and quality of B cell and antibody responses to pertussis immunization with the TDaP vaccine.
2. Assess the impact of HIV infection and of the timing of maternal immunization on the transplacental transfer and on the quality of pertussis-specific IgG in the newborn.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* HIV-infected or uninfected pregnant women in their second/third trimester with an indication of TDaP vaccination
* Non pregnant HIV negative women (having a negative HIV test in the last 6 months or at screening) with an indication of TDaP vaccination

Exclusion Criteria:

* Grade III/IV anemia
* Active bacterial infection
* Opportunistic infection (Tuberculosis, CMV, toxoplasmosis, etc)
* Inability to understand the nature and extent of the study and the procedures required
* Current or recent use of immunosuppressive drugs (corticosteroids, anti-TNF, methotrexate, etc)
* Active neoplasia

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnancy
Study Population: Recruitment at the Pre-natal clinic for pregnant women (HIV-infected or uninfected) on voluntary basis Recruitment at the Travel & Vaccine Clinic for HIV-uninfected non-pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Pertussis-specific antibodies GMC after immunization | 7-10 days, 30 days and at delivery for pregnant women
  Anti-Pertussis Toxin (PT), Filamentous Hemagglutinin (FHA) and pertactin (PRN) specific antibodies levels
Transplacental transfer of pertussis-specific antibodies | Birth
  Anti-PT, FHA and PRN specific antibodies levels transfer ratio

SECONDARY OUTCOMES:
Pertussis-specific memory B cells quantification & phenotype | 7-10 days, 30 days and at delivery for pregnant women
  PT, FHA and PRN-specific memory B cells numbers assessed by ELISPOT assay & Flow Cytometry
Pertussis-specific antibodies glycosylation profiles | 7-10 days, 30 days and at delivery for pregnant women
  Anti-PT, FHA and PRN specific antibodies profiles

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Dauby, M.D. Ph.D., Principal Investigator — Centre Hospitalier Universitaire Saint Pierre
Locations (2):
- Belgium (2):
  - CHU Saint-Pierre, Brussels
  - HIS Etterbeek Ixelles, Ixelles-Elsene

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Taton M, Willems F, Widomski C, Martin C, Jiang Y, Renard K, Cogan A, Necsoi C, Ackerman ME, Marchant A, Dauby N. Impact of pregnancy on polyfunctional IgG and memory B cell responses to Tdap immunization. Vaccine. 2023 Jun 19;41(27):4009-4018. doi: 10.1016/j.vaccine.2023.05.035. Epub 2023 May 25. PMID 37244810